CLINICAL TRIAL: NCT04928625
Title: An Open-Label, Single-Arm, Multi-Center Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-A1904 in Patients With Advanced Pancreatic Cancer
Brief Title: A Trial of SHR-A1904 in Patients With Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1904-I-102
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-05

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Intervention Model Description: Open-Label, Single-Arm, Multi-Center Phase I Clinical Study TO EVALUATE the Safety
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1904 (Experimental)
  Interventions: Drug: SHR-A1904

INTERVENTIONS:
Drug: SHR-A1904 — SHR-A1904

SUMMARY:
The study is being conducted to assess the safety and tolerability of SHR-A1904 in patients with with advanced pancreatic cancer and to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and recommended phase II dose (RP2D) of SHR-A1904

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
2. Males or females aged 18-75 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Has a life expectancy of ≥ 3 months
5. Has at least one measurable lesion as defined by RECIST v1.1

Exclusion Criteria:

1. Plan to receive any other anti-tumor treatments during the study treatment period of this study
2. Received other clinical investigational products or treatments within 4 weeks before the first dose of the study
3. Underwent a major surgery other than diagnosis or biopsy within 4 weeks before the first dose of the study
4. Previously received gastrectomy (only for subjects of the dose-escalation part)
5. Subjects with known brain metastases
6. Grade II-IV cardiac insufficiency as per the New York Heart Association (NYHA) criteria; arrhythmia requiring long-term drug control; unstable angina or acute myocardial infarction within 6 months before the first dose of the study
7. Presence of accompanying diseases (such as poorly controlled hypertension, serious diabetes mellitus, thyroid disorder, psychosis, etc.) that may pose serious risks to the safety of the subject or may affect the subject's ability to complete the study, or any other situation as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of SHR-A1904 | UP to 2 months
Maximum tolerated dose (MTD) of SHR-A1904 | UP to 2 months
Recommended Phase II Dose (RP2D) | Up to 1 year

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 1 year
Time to maximum concentration (Tmax) | up to 1 year
Area under the drug concentration-time curve from time 0 to the last measurable concentration time point (AUC0-t) | Up to 1 year
Anti-drug antibody (ADA) of SHR-A1904 | Up to 1 year
Objective response rate (ORR) | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China